CLINICAL TRIAL: NCT00003422
Title: A Randomised Trial Comparing Pre-Operative Radiotherapy and Selective Post-Operative Chemoradiotherapy in Rectal Cancer
Brief Title: Radiation Therapy Before Surgery Compared With Chemotherapy Plus Radiation After Surgery in Treating Patients With Rectal Cancer That Can Be Surgically Removed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Collaborators: NCIC Clinical Trials Group (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066442; MRC-CR07; EU-98008; CAN-NCIC-C016; ISRCTN28785842
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2007-03

CONDITIONS: Colorectal Cancer
Keywords: stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether giving radiation therapy before surgery is more effective than giving chemotherapy plus radiation therapy after surgery in treating patients with rectal cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy given before surgery to see how well it works compared to chemotherapy and radiation therapy given after surgery in treating patients with rectal cancer that can be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare local recurrence free rates and quality of life in patients with operable rectal cancer receiving preoperative radiotherapy versus patients receiving selective postoperative chemoradiotherapy.
* Determine local recurrence free survival, overall survival, time to appearance of distant metastases, disease free survival and morbidity in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by a number of factors including surgeon.

Patients are randomized to receive preoperative radiotherapy (arm I) or postoperative chemoradiotherapy (arm II).

* Arm I: Patients receive radiotherapy in 5 fractions over 1 week prior to surgery. Patients undergo surgery within 7 days of the last fraction of radiotherapy.
* Arm II: Patients receive chemoradiotherapy 4-12 weeks after surgery (if circumferential resection margins are histologically involved by tumor). Radiotherapy is administered in 25 fractions over 5 weeks (5 days per week). During radiotherapy, patients either receive fluorouracil (5-FU) continuous infusion, 5-FU bolus IV and leucovorin calcium IV weekly, or a 5-day bolus schedule of 5-FU and leucovorin calcium.

Patients may then receive adjuvant chemotherapy as per local policy.

Quality of life assessments are made every 3 months for 1 year and then every 6 months for the next 2 years.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 1800 patients will be accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum (defined as lower edge of tumor within 15 cm of anal verge)
* Tumor considered potentially operable
* No evidence of metastases indicated by liver ultrasound or CT scan; chest x-ray; or renal, liver, and bone profiles

PATIENT CHARACTERISTICS:

Age:

* 75 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No uncontrolled heart failure or angina

Other:

* No other concurrent uncontrolled medical illness (e.g., infection)
* No other prior or concurrent malignancy likely to interfere with the protocol treatments or comparisons

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 1998-01; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Local recurrence by biopsy, imaging, or imaging and carcinoembryonic antigen result

SECONDARY OUTCOMES:
Local recurrence-free survival
Overall survival
Time to appearance of distant metastases
Disease-free survival
Morbidity
Quality of life
Economic implications

CONTACTS AND LOCATIONS:
Overall Officials: R. Steele, Study Chair — Ninewells Hospital; Jean Couture, MD, Study Chair — Hopital Charles Lemoyne
Locations (9):
- Canada (8):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - St. Catharines General Hospital at Niagara Health System, St. Catharines, Ontario
  - Toronto Sunnybrook Regional Cancer Centre at Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
- Ninewells Hospital and Medical School, Dundee, Scotland, United Kingdom

REFERENCES:
- [Result] Stephens RJ, Thompson LC, Quirke P, Steele R, Grieve R, Couture J, Griffiths GO, Sebag-Montefiore D. Impact of short-course preoperative radiotherapy for rectal cancer on patients' quality of life: data from the Medical Research Council CR07/National Cancer Institute of Canada Clinical Trials Group C016 randomized clinical trial. J Clin Oncol. 2010 Sep 20;28(27):4233-9. doi: 10.1200/JCO.2009.26.5264. Epub 2010 Jun 28. PMID 20585099
- [Result] Quirke P, Steele R, Monson J, Grieve R, Khanna S, Couture J, O'Callaghan C, Myint AS, Bessell E, Thompson LC, Parmar M, Stephens RJ, Sebag-Montefiore D; MRC CR07/NCIC-CTG CO16 Trial Investigators; NCRI Colorectal Cancer Study Group. Effect of the plane of surgery achieved on local recurrence in patients with operable rectal cancer: a prospective study using data from the MRC CR07 and NCIC-CTG CO16 randomised clinical trial. Lancet. 2009 Mar 7;373(9666):821-8. doi: 10.1016/S0140-6736(09)60485-2. PMID 19269520
- [Result] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S, Quirke P, Couture J, de Metz C, Myint AS, Bessell E, Griffiths G, Thompson LC, Parmar M. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet. 2009 Mar 7;373(9666):811-20. doi: 10.1016/S0140-6736(09)60484-0. PMID 19269519
- [Result] Quirke P, Sebag-Montefiore D, Steele R, et al.: Local recurrence after rectal cancer resection is strongly related to the plane of surgical dissection and is further reduced by pre-operative short course radiotherapy. Preliminary results of the Medical Research Council (MRC) CR07 trial. [Abstract] J Clin Oncol 24 (Suppl 18): A-3512, 2006.
- [Result] Sebag-Montefiore D, Steele R, Quirke P, et al.: Routine short course pre-op radiotherapy or selective post-op chemoradiotherapy for resectable rectal cancer? Preliminary results of the MRC CR07 randomised trial. [Abstract] J Clin Oncol 24 (Suppl 18): A-3511, 2006.
- [Result] Sebag-Montefiore D: An update report on the MRC CR07 trial. [Abstract] Br J Cancer 85 (suppl 1): A-9.3, 28, 2001.